CLINICAL TRIAL: NCT05856370
Title: The Ailliance Post-Market Clinical Study: All enablIng technoLogies, bioLogics, IDS, And Core spiNe produCt collEction
Brief Title: The Ailliance Post-Market Clinical Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Spinal and Biologics (Industry)
Collaborators: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: MDT22045CSTAIL
Record Dates: First submitted 2023-03-16; First posted 2023-05-12 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Spinal Deformity; Spinal Degenerative Disorder; Spinal Fusion Failure; Spinal Trauma; Spinal Tumor Case

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Receiving eligible Medtronic device(s) from all product groups (Other): Powered Systems, Instruments, and Imaging device(s), Advanced Energy device(s), Robotics and Navigation, Rods and Screws, Interbodies and Biologics, Spinal Tethers, and Other Spinal Hardware device(s)
  Interventions: Device: Follow-up schedule: pre-operative baseline up to 24-months post-procedure

INTERVENTIONS:
Device: Follow-up schedule: pre-operative baseline up to 24-months post-procedure — Follow-up assessments will be required (therefore interventional) from pre-operative baseline to 24 months post index surgery

SUMMARY:
The purpose of this clinical study is to collect performance and safety data for post-market Medtronic devices indicated for cranial and/or spinal indication(s).

Subjects are enrolled and followed postoperatively to 24 months. The Ailliance clinical study is intended to collect data congruous with routine clinical care practices.

ELIGIBILITY:
Inclusion Criteria:

1. Subject provides written informed consent per institution and/or geographical requirements.
2. Subject is intended to receive or be treated with an eligible Medtronic Cranial and Spinal Technology (CST) device(s) (see product appendices), used alone or in combination, for a cranial and/or spinal indication(s).
3. Subject is at least 18 years of age or minimum legal age as required by local regulations.
4. Subject agrees to complete all required assessments per the Schedule of Events.

Exclusion Criteria:

1. Subject is currently enrolled or plans to enroll in concurrent drug/device/biologic trial(s) that may confound this trial's results per investigator assessment (i.e. no required intervention that could affect interpretation of all-around device safety and or performance).
2. Subject who is, or is expected to be, inaccessible for all required follow-up visits.
3. Subject with exclusion criteria required by local law.
4. Subject is considered vulnerable at the time of obtaining consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2031-05 (Estimated); Study Completion 2031-05 (Estimated)

PRIMARY OUTCOMES:
Surgical success (for any Medtronic eligible market-released Advanced Energy device(s) used) | Discharge (from Index Surgery completion to 14 days post-operatively)
  Defined by amount of: 1) blood loss (mL) during surgery and/or 2) total operation time and/or 3) length of stay in the hospital (measured from surgery completion to discharge), and/or 4) investigator opinion on whether the device(s) directly assisted in the completion of surgery
Fusion Success (for any Medtronic eligible market-released Interbodies and Biologics, Other Spinal Hardware, and/or Rods and Screws device(s) used) | 12 months
  Fusion success at 12-months is determined through evaluation of radiographic evidence (X-ray and/or CT scan) by the investigator by: (1) Confirming the presence of bone bridging, and (2) if using the Brantigan & Steffee's Classification scale: a score D and/or E are determined.
Surgical performance (for any Medtronic eligible market-released Powered Systems, Instruments, and Imaging device(s) used) | Index Surgery
  Surgical performance, as defined as the rate at which the device directly assisted in the completion of surgery in the investigator's opinion.
  If O-Arm used: whether O-Arm was utilized for validation of implant placement during the surgery.
Device performance (for any Medtronic eligible market-released Robotics and Navigation device(s) used) | 24 months
  Robotics: Planned number of screws prior to index surgery compared to number of screws device assisted with placement during surgery. Navigation: Whether or not device was utilized for validation of screw placement during surgery.
Pain Resolution (for select Medtronic eligible market-released Other Spinal Hardware device(s) used) | 12 months
  Resolution of pain at 12-months when compared to baseline Pain reported by the subject using the Neck Disability Index (NDI) questionnaire
Stabilization (for any Medtronic eligible market-released device(s) used from the following product groups: Other Spinal Hardware) | Up to 12 months
  * Stabilization is the radiographic verification of no noticeable hardware and/or implant loosening, the presence of the hardware in the appropriate position without cage subsidence and/or implant loosening, and noticeable stable alignment of the spine post-surgery.
  * Since all products are market-released, assessment for stabilization will be completed by the investigator.
  * Stabilization will be assessed by the collection of radiographic evidence (X-Ray(s) and CT-scan(s)).
Deformity Correction (for specified Medtronic eligible market-released device(s) used from the following product groups: Spinal Tethers) | 12 months
  Defined by the change of Cobb angle at 12-month

SECONDARY OUTCOMES:
Rate of Device-related Adverse Events any Medtronic eligible market-released Cranial & Spinal Technologies (CST) device(s) as aligned with ISO 14155 standards | 24 months
  The secondary endpoint is defined as the rate of occurrence for device-related adverse events
Stabilization [for any Medtronic eligible market-released device(s) used from the following product groups: Interbodies and Biologics, Rods and Screws] | Up to 12 months
  * Stabilization is the radiographic verification of no noticeable hardware and/or implant loosening, the presence of the hardware in the appropriate position without cage subsidence and/or implant loosening, and noticeable stable alignment of the spine post-surgery.
  * Since all products are market-released, assessment for stabilization will be completed by the investigator.
  * Stabilization will be assessed by the collection of radiographic evidence (X-Ray(s) and CT-scan(s)).
Deformity Correction [for specified Medtronic eligible market-released device(s) used from the following product groups: Rods and Screws] | 12 months
  * Deformity correction is defined by the change of Cobb angle at the 12-month postoperative visit compared to baseline.
  * Assessment(s) for deformity correction will be completed by the investigator. The investigator will determine whether the subject meets requirements of deformity correction based on the comparison of the Cobb angle measurements at all postoperative visits, when compared to the subject's baseline assessments.
  * Cobb angle measurements will be provided through collection of radiographic evidence (X-Ray(s) and CT-scan(s)) and assessed by the investigator.

CONTACTS AND LOCATIONS:
Locations (23):
- United States (20):
  - University of Arizona, Tucson, Arizona
  - OrthoArkansas, Little Rock, Arkansas
  - University of California Davis Medical Center, Sacramento, California
  - University of California, San Francisco (UCSF), San Francisco, California
  - Indiana University School of Medicine, Bloomington, Indiana
  - Indiana Spine Group, Carmel, Indiana
  - The Orthopaedic Research Foundation (OrthoIndy), Indianapolis, Indiana
  - Norton Leatherman Spine Specialists, Louisville, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - Michigan Orthopaedic & Spine Surgeons, Rochester Hills, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University at Buffalo, Buffalo, New York
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Pittsburgh Medical Center UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Rhode Island Hospital University Orthopedic, Providence, Rhode Island
  - Tennessee Orthopaedic Alliance, Nashville, Tennessee
  - American Neurospine Institute, PLLC, Frisco, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Virginia Spine Institute, Reston, Virginia
- Hôpital Roger Salengro, Lille, France
- Hospital Vall D'Hebron, Barcelona, Spain
- Kings College Hospital NHS Foundation Trust, London, United Kingdom